CLINICAL TRIAL: NCT05525819
Title: The Effect of Intrathecal Versus Intravenous Dexmedetomidine on Postoperative Analgesia in Transurethral Resection of The Prostate
Brief Title: Intrathecal Versus Intravenous Dexmedetomidine in Prostate Transurethral Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Laila Elahwal, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 34141/9/20
Record Dates: First submitted 2022-08-29; First posted 2022-09-02 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Dexmedetomidine; Transurethral Resection of Prostate; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): Cases will be subjected to spinal anesthesia with hyperbaric bupivacaine 10 mg.
  Interventions: Drug: Control group
- Intrathecal group (Experimental): Cases will be subjected to the same anesthetic mixture as controls with adding dexmedetomidine 5 μg.
  Interventions: Drug: Intrathecal group
- Intravenous group (Experimental): Cases will receive hyperbaric bupivacaine (10 mg), in addition to IV dexmedetomidine (1 μg/kg loading dose, followed by 0.4 μg/kg/h maintenance dose).
  Interventions: Drug: Intravenous group

INTERVENTIONS:
Drug: Control group — The cases will be subjected to spinal anesthesia with a 3 ml volume (2.5 ml of hyperbaric bupivacaine 10 mg in addition to 0.5 normal saline). 50 ml of normal saline was infused over a ten-minute period, followed by 200 ml infusion till the end of operation.
  Arms: Control group
Drug: Intrathecal group — The cases will be subjected to the same anesthetic mixture as controls with adding dexmedetomidine 5 μg in the saline component. 50 ml of normal saline was infused over a ten-minute period, followed by 200 ml infusion till the end of operation.
  Arms: Intrathecal group
Drug: Intravenous group — The intravenous group will receive 2.5 ml of hyperbaric bupivacaine (10 mg), in addition to intravenous dexmedetomidine, which will be started at 1 μg/kg loading dose diluted in 50 ml saline administered within 10 min, followed by maintenance at a 0.4 μg/kg/h dose diluted in 200 ml saline till the end of the procedure.
  Arms: Intravenous group

SUMMARY:
This study was conducted to compare the effects of intrathecal versus intravenous dexmedetomidine administration in patients undergoing Transurethral resection of the prostate under spinal anesthesia.

DETAILED DESCRIPTION:
Multiple prostatic pathologies become evident in the elderly males. Of them, benign prostatic hyperplasia is one of the most prevalent issues in aging men and transurethral resection of the prostate (TURP) still represents the standard surgical treatment.

Most transurethral resection of the prostate (TURP) procedures are performed under spinal anesthesia. Spinal anesthesia has many advantages including, easy application, low cost, decreasing the risk of aspiration, decreasing intraoperative bleeding, eliminating the need for mechanical ventilation together with the decreased risk of intraoperative cardiac events or post-operative hypoxic episode.

The management of post-operative pain following spinal anesthesia using a short-acting anesthetic still constitutes a major problem for anesthesiologists and pain physicians. However, the duration and efficacy of spinal anesthesia could be improved by adjuvants.

Dexmedetomidine is an alpha 2 receptor agonist that have antinociceptive action for both visceral and somatic pain. At low doses, it has sedative and hypnotic effects without having a negative impact on respiration. Multiple studies have reported that intrathecal and intravenous administration of this drug could prolong the duration of spinal anesthesia and post-operative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Cases aged between 50 and 70 years
* Having class I or II according to the American society of anesthesiologists (ASA)

Exclusion Criteria:

* Cases with heart block
* Dysrhythmia
* Contraindications for spinal anesthesia
* Known allergy to the study medications
* Classified as ASA class > II
* Alpha 2 agonist or antagonist therapy.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-29 (Estimated); Study Completion 2023-04-29 (Estimated)

PRIMARY OUTCOMES:
Time to first analgesic request | 24 hours postoperatively
  Time to first analgesic request will be recorded

SECONDARY OUTCOMES:
The onset of sensory | 24 hours Postoperatively
  Time to reach T7 sensory block will be recorded
The degree of motor block | 24 hours Postoperatively
  The degree of motor block will be assessed using the modified Bromage Score. Grade 0 No motor block Grade 1 Inability to raise extended leg, able to move knees and feet Grade 2 Inability to raise extended leg and move knee, able to move feet Grade 3 Complete motor block of the lower limbs.
Sedation level | Intraoperativley
  Patients level of sedation will be assessed via Ramsay sedation score. This score is numbered from 1 to 6, based on patient responsiveness.
Total analgesic requirements | 48 hours Postoperatively
  Total analgesic requirements will be recorded
The incidence of side effects | 48 hours Postoperatively
  The incidence of side effects including (bradycardia, hypotension, nausea, vomiting, and pruritis) will be recorded..

CONTACTS AND LOCATIONS:
Locations (1):
- Surgical Intensive Care and Pain Medicine Department, Faculty of Medicine, Tanta University, Tanta, Egypt, Tanta, ElGharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All information will be available under a reasonable request from the corresponding author
Supporting Information: Study Protocol
Time Frame: One year after the completion of the study